CLINICAL TRIAL: NCT06290076
Title: A Predictive Model and Scoring System for Severe Complications After Endovascular Thrombectomy: a Retrospective, Multicenter, Observational Study
Brief Title: A Predictive Model and Scoring System for Severe Complications After Endovascular Thrombectomy
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: IAT-PROACT
Record Dates: First submitted 2024-02-07; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke; Endovascular Thrombectomy; Symptomatic Intracranial Hemorrhage; Malignant Cerebral Edema
Keywords: Acute Ischemic Stroke; Endovascular Thrombectomy; sICH; MCE
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe Complications Group: Patients with severe complications (including symptomatic intracranial hemorrhage and malignant cerebral edema) occurred within 72 hours after endovascular thrombectomy are classified into severe complications group.
- Non-Severe Complications Group: Patients without severe complications (including symptomatic intracranial hemorrhage and malignant cerebral edema) occurred within 72 hours after endovascular thrombectomy are classified into non-severe complications group.

SUMMARY:
To establish a predictive model and scoring system for predicting severe complications after thrombectomy. This scoring system can be used to identify high-risk patients after endovascular thrombectomy, guide the early use of adjunctive interventions, and provide reference for future clinical trials.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) accounts for about 80% of all strokes. The focus of AIS treatment is to restore reperfusion of ischemic territory as soon as possible, promote neurological recovery, reduce disability rate and improve long-term survival rate. In recent years, a series of randomized clinical trials have proved that endovascular thrombectomy (EVT) is safe and effective in the treatment of anterior circulation AIS. EVT has been recommend as the first-line treatment for anterior circulation large vessel occlusion (LVO) stroke by guidelines.

Symptomatic intracranial hemorrhage (sICH) and malignant cerebral edema (MCE) are the two most common severe neurological complications, leading to brain tissue hypoxia and neurological dysfunction. Currently, there is a lack of prediction system to identify patients at high risk for severe complications, who can most likely benefit from adjuvant treatment after thrombectomy to improve patient functional independence and survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms and signs compatible with ischemia in the anterior circulation
2. Internal carotid artery occlusion or middle cerebral artery M1 and M2 segment occlusion confirmed by computed tomographic angiography (CTA)/ magnetic resonance angiography (MRA)/ digital subtraction angiography (DSA)
3. Premorbid mRS ≤1;
4. National Institutes of Health Stroke Score (NIHSS) ≥6 at admission;
5. Onset to puncture time ≤24h;
6. Treated with thrombectomy resulting in mTICI score ≥2b at end of the procedure.

Exclusion Criteria:

1. Intracranial hemorrhage, aneurysm, and arteriovenous malformation before endovascular thrombectomy;
2. Perioperative complications, including dissection and arterial perforation;
3. Anticipated life expectancy <3 months;
4. Critical baseline clinical, laboratory and imaging data are missing;
5. Lack of follow-up results within 72 hours and 90 days after thrombectomy;
6. Pregnant or lactating women;
7. Severe systemic diseases (e.g. advanced cancer), potentially interfering with prognosis;
8. Allergy to contrast media and nitinol;
9. Concurrent participation in a study that would interfere with the establishment of predictive models;
10. Unable to complete the assessment due to mental disorders cognitive or emotional disorders before onset.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At least 1500 patients with anterior circulation acute ischemic stroke due to large vessel occlusion and received endovascular thrombectomy.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of severe complications | Within 72 hours after thrombectomy
  Severe complications include symptomatic intracranial hemorrhage (sICH) and malignant cerebral edema (MCE). SICH was defined as any intracranial hemorrhage on the non-contrast CT scan accompanied with clinical deterioration, as defined by a increase of ≥4 points in the NIHSS score, or that led to death and that was identified as the predominant cause of the neurologic deterioration.
  MCE was defined as a malignant state in which neurological function deteriorates progressively due to brain edema after endovascular thrombectomy, causing disturbance of consciousness, anisocoria, and midline shift of 5 mm or more on imaging, leading to brain herniation or death. Midline shift was obtained by measuring the point of maximum deviation perpendicular to the line connecting the anterior and posterior attachment points of the falx cerebri.

SECONDARY OUTCOMES:
Rate of mRS score of 3-6 | 90 days (±7 days) after thrombectomy
  The mRS score range from 0 (no disability) to 6 (death)
Rate of mRS score of 5-6 | 90 days (±7 days) after thrombectomy
  The mRS score range from 0 (no disability) to 6 (death)
Rate of symptomatic intracranial hemorrhage | Within 72 hours after thrombectomy
  SICH was defined as any intracranial hemorrhage on the non-contrast CT scan accompanied with clinical deterioration, as defined by a increase of ≥4 points in the NIHSS score, or that led to death and that was identified as the predominant cause of the neurologic deterioration.
Rate of malignant cerebral edema | Within 72 hours after thrombectomy
  MCE was defined as a malignant state in which neurological function deteriorates progressively due to brain edema after endovascular thrombectomy, causing disturbance of consciousness, anisocoria, and midline shift of 5 mm or more on imaging, leading to brain herniation or death. Midline shift was obtained by measuring the point of maximum deviation perpendicular to the line connecting the anterior and posterior attachment points of the falx cerebri.
Change of NIHSS score | 24-72 hours after thrombectomy versus admission
  The NIHSS score range from 0 (no deficit) to 42 (maximum deficit)
Rate of modified Rankin Scale (mRS) score of 0-2 | 90 days (±7 days) after thrombectomy
  The mRS score range from 0 (no disability) to 6 (death)
All-cause mortality | 90 days (±7 days) after thrombectomy
  Death defined as a mRS score of 6

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Z, Hao J, Wen C, Cheng T, Zhao Y, Bai X, Guo X, Cao W, Li T, Min XL, Jiao L, Zhang L, Yang B. Predictive factors for very poor outcomes after endovascular thrombectomy in anterior circulation large vessel occlusion: a multicentre retrospective study in China. BMJ Open. 2025 Oct 23;15(10):e101244. doi: 10.1136/bmjopen-2025-101244. PMID 41130675